CLINICAL TRIAL: NCT03488225
Title: Phase II Study of the Hyper-CVAD Regimen in Sequential Combination With Inotuzumab Ozogamicin as Frontline Therapy for Adults With B-Cell Lineage Acute Lymphocytic Leukemia
Brief Title: Combination Chemotherapy and Inotuzumab Ozogamicin in Treating Patients With B Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the study was closed early due to competing trials
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0922; NCI-2018-00760 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0922 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-04-04 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia in Remission; B Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Inotuzumab Ozogamicin; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; ofatumumab; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (hyper-CVAD, inotuzumab ozogamicin) (Experimental): See detailed description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Biological: Inotuzumab Ozogamicin; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Biological: Ofatumumab; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; BW 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, IV or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well combination chemotherapy and inotuzumab ozogamicin work in treating patients with B acute lymphoblastic leukemia. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, dexamethasone, methotrexate and cytarabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as inotuzumab ozogamicin, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving combination chemotherapy and inotuzumab ozogamicin may work better at treating B acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical efficacy of the sequential combination of hyper-CVAD (hyperfractionated cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, dexamethasone, methotrexate and cytarabine) + inotuzumab ozogamicin in patients with newly diagnosed B-cell acute lymphocytic leukemia (ALL) in terms of event-free survival (EFS).

SECONDARY OBJECTIVES:

I. To evaluate other efficacy endpoints such as overall survival, overall response rate, minimal residual disease (MRD) negativity rate as well as the safety of this combination.

OUTLINE:

INTENSIVE CHEMOTHERAPY: Patients receive cyclophosphamide intravenously (IV) over 3 hours every 12 hours on days 1-3 and dexamethasone IV or orally (PO) on days 1-4 and 11-14 of courses 1 and 3. Patients may receive ofatumumab IV over 2 hours on days 1, 2 and 11 of course 1, days 1 and 8 of courses 2 and 4, and days 1 and 11 of course 3, or rituximab IV over 2 hours on days 1 and 11 of courses 1 and 3, and days 1 and 8 of courses 2 and 4. Patients also receive methotrexate intrathecally (IT) on day 2 of courses 1 and 3, IV over 24 hours on day 1 and IT on day 8 of courses 2 and 4, doxorubicin hydrochloride IV over 24 hours on day 4 of courses 1 and 3, vincristine sulfate IV over 1 hour on days 4 and 11 of courses 1 and 3, cytarabine IT on day 7 of courses 1 and 3, and IV over 2 hours every 12 hours on days 2 and 3, and IT on day 5 of courses 2 and 4, leucovorin calcium IV 4 times a days on day 2 of courses 2 and 4. Patients then receive inotuzumab ozogamicin IV over 1 hour on days 1 and 8 of courses 5-8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive mercaptopurine PO thrice a day, methotrexate PO once a week, vincristine sulfate IV over 1 hour on day 1 and prednisone PO on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, previously untreated B-lineage ALL, or having achieved complete remission (CR) with one course of induction chemotherapy
* Patients with extramedullary disease only are eligible
* Failure to one induction course of chemotherapy (these patients will be analyzed separately)
* Performance status of 0-3
* Creatinine less than or equal to 2.0 mg/dL (unless considered tumor related)
* Bilirubin less than or equal to 2.0 mg/dL (unless considered tumor related)
* Adequate cardiac function as assessed by history and physical examination
* No active or co-existing malignancy with life expectancy less than 12 months
* Women of childbearing potential (WOCBP) or male subjects with a partner who is WOCBP must agree to use contraception during the study, if sexually active

Exclusion Criteria:

* Pregnant or nursing women
* Known to be human immunodeficiency virus (HIV)-positive
* Philadelphia chromosome (Ph)-positive ALL
* Active and uncontrolled disease/infection as judged by the treating physician
* Unable or unwilling to sign the consent form
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver involvement or stable chronic liver disease per investigator assessment)
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active hepatitis C

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2018 to January 2019
Period: Overall Study
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Off Protocol Therapy | 2
Not completed — Stem Cell Transplant | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 29 [19 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival
Description: Event-free survival defined as the time interval from date of treatment start until the date of death, disease progression or relapse.
Time Frame: Start of treatment up to 2 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Months | 24 [18.5 to 24]

2. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Start of treatment up to 2 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Months | 24 [18.5 to 24]

3. Secondary Outcome: Participants to Achieve Complete Remission (CR):
Description: Complete Remission (CR) is defined as - Normalization of the peripheral blood and bone marrow blasts </= 5% in normocellular or hypercellular marrow, granulocyte count of 1x10^9/L or above and platelets >/= 100X10^9/L and complete resolution of all sites of extramedullary disease.
Time Frame: Start of treatment up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Participants | 4

4. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD) Negativity
Description: MRD levels continuously assessed during induction and consolidation therapy by 6-color multiparameter flow. MRD negativity defined by a value of at least 10-4 and confirmed on a second bone marrow aspiration/biopsy performed after a subsequent cycle.
Time Frame: Start of treatment up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Number of Participants With Adverse Events
Description: For the purpose of toxicity monitoring, toxicities are defined as any treatment -related grade 3 or 4 non-hematologic AEs occurred any time during the trial.NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 utilized for adverse event reporting.
Time Frame: Start of treatment up to 30 days after last dose received.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
Number analyzed (Participants) | 4
Participants
  Neutropenic Fever | 2
  Peripheral Sensory Neuropathy | 1
  Allergic Reaction | 1
  Muscle Weakness | 1

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin) (N=4)
Neutropenic Fever (Blood and lymphatic system disorders) | 2 (2)
Kidney Infection (Infections and infestations) | 1 (1)
Fever (General disorders) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hyper-CVAD, Inotuzumab Ozogamicin) (N=4)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 2 (3)
Allergic Reaction (Immune system disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema Limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Infusion Related Reaction (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutropenia (Investigations) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Oral Mucositis (Gastrointestinal disorders) | 3 (4)
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (4)
Sinus Bradycardia (Cardiac disorders) | 2 (2)
Thrombocytopenia (Investigations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (2)
Arachnoiditis (Nervous system disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03488225/Prot_SAP_000.pdf